CLINICAL TRIAL: NCT02079818
Title: CLP 7463: Visceral Artery Aneurysm Embolization by the Penumbra Ruby™ Coil System
Brief Title: Visceral Artery Aneurysm Embolization by the Penumbra Ruby™ Coil System
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was never initiated.
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP 7463
Record Dates: First submitted 2014-03-03; First posted 2014-03-06 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Visceral Artery Aneurysms; Arteriovenous Malformations
Keywords: visceral artery aneurysms; arteriovenous malformations; Penumbra Ruby Coil System
MeSH Terms: conditions — Arteriovenous Malformations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Penumbra Ruby Coil System (Experimental)
  Interventions: Device: Penumbra Ruby Coil System

INTERVENTIONS:
Device: Penumbra Ruby Coil System — The Penumbra Ruby™ Coil is a new generation of detachable coils developed by Penumbra Inc. This coil system is specifically designed for the occlusion of aneurysms and vessels that is equivalent to standard platinum coils. This system consists of: an implantable Coil attached to a Detachment Pusher as well as a Detachment Handle. The Detachment Pusher is comprised of a shaft with a radiopaque positioning marker, a Distal Detachment Tip, and a pull wire. The Detachment Handle is used to detach the Coil Implant from the Detachment Pusher. The Penumbra Ruby Coil is designed for endovascular embolization in the peripheral vasculature. Intended users for this device are physicians who have received appropriate training in interventional radiology and endovascular intervention.

SUMMARY:
The primary objective of this study is to gather post market data on the Penumbra Ruby Coil System in the treatment of visceral artery aneurysms and arteriovenous malformations. This study is a prospective, multi-center study of patients with visceral artery aneurysms and visceral arteriovenous malformations who are treated by the Penumbra Ruby Coil System. Data for each patient are collected up to 12 months post-procedure for the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in this study must be those treated according to the cleared indication for the Penumbra Ruby Coil System for visceral arterial and venous embolizations.

Exclusion Criteria:

* Patients in whom endovascular embolization therapies other than Penumbra Coils are used will be excluded from this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
1. Packing density with the number of coils implanted | During the procedure
2. Time of fluoroscopic exposure | During the procedure
3. Procedural device-related serious adverse events at immediate post-procedure | At immediate post-procedure
4. Occlusion of the aneurysm sac or target vessel at immediate post-procedure | At immediate post-procedure
5. Occlusion of the aneurysm sac or target vessel at one year post-procedure | One year post-procedure

SECONDARY OUTCOMES:
1. Recanalization of the aneurysm sac or target vessel at 4 months post-procedure | 4 months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Paraq J Patel, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States